CLINICAL TRIAL: NCT01269541
Title: MESS- MRSA Eradication Study Skåne. A Comparison Between Systemic Antibiotic Treatment in Combination With Topical Mupirocintreatment With Only Topical Mupiroicintreatment to Eradicate MRSA in Throat Carriers
Brief Title: MESS-study MRSA Eradication Study Skåne
Acronym: MESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRSA-2010; 2010-019727-55 (EudraCT Number)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2015-05

CONDITIONS: Throatcarriers of MRSA
MeSH Terms: interventions — Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mupirocin (Active Comparator): Topical treatment
  Interventions: Drug: Mupirocin; Drug: Rifampin+Clindamycine or Trimehoprimsulfa
- Rifampicin+Clindamycine or Trimethoprimsulfa (Active Comparator): Rifampicin 10 mg/kgx1xVII Clindamycine 300 mgx3xVII Trimethoprimsulfa 400mg/80mg 2x2
  Interventions: Drug: Rifampin+Clindamycine or Trimehoprimsulfa

INTERVENTIONS:
Drug: Mupirocin — Topical in the nose 3 times daily for 5 days
  Arms: Mupirocin
Drug: Rifampin+Clindamycine or Trimehoprimsulfa — Rifampicin 10 mg/kgx1xVII Clindamycine 300 mgx3 Trimethoprimsulfa 400mg/80mg 2x2

SUMMARY:
The purpose of this study is to determine whether systemic antibiotic treatment with rifampicin and clindamycine or trimethoprim-sulfa in addition to topical treatment with mupirocin is more effective than only topical treatment to eradicate MRSA in throatcarriers

ELIGIBILITY:
Inclusion Criteria:

Colonized with MRSA in the throat Older than 5 years MRSA-bacteria sensitive for Rifampicin and Clindamycine or Trimethoprimsulfa -

Exclusion Criteria:

Allergy to the studymedication Healthcareworkers Pregnancy Active infection with MRSA Immunosuppression Treatment with other antibiotic during the studyperiod

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Culture for MRSA | after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Melander, MD PHD, Principal Investigator — Labmedicin Skåne Malmö
Locations (6):
- Sweden (6):
  - Helsingborg hospital, Helsingborg, Skåne County
  - Kristianstad hospital, Kristianstad, Skåne County
  - Infectious department SUS Lund, Lund, Skåne County
  - SUS Malmö, Malmo, Skåne County
  - Örebro university hospital, Örebro
  - Karolinska university hospital, Stockholm